CLINICAL TRIAL: NCT04527432
Title: A Pilot Assessment of the COVID-19 Antibody Status and Associated Factors, in Individuals Employed by a Large Acute NHS Trust During the Coronavirus Pandemic
Brief Title: COVID-19 Health Professional Impact Study
Acronym: CHIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Royal Wolverhampton Hospitals NHS Trust (Other Government)
Collaborators: University of Wolverhampton (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2020COV112
Record Dates: First submitted 2020-08-24; First posted 2020-08-26 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-04

CONDITIONS: Coronavirus Infection; Severe Acute Respiratory Syndrome
MeSH Terms: conditions — Coronavirus Infections; Severe Acute Respiratory Syndrome | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All participants (Other): Survey at 6 and 12 months time with optional antibody tests
  Interventions: Other: Survey; Diagnostic Test: SARS-CoV-2 antibody test

INTERVENTIONS:
Other: Survey — Survey at baseline, 6 and 12 months
Diagnostic Test: SARS-CoV-2 antibody test — SARS-CoV-2 antibody test results and testing again at 6 and 12 months

SUMMARY:
The COVID-19 (coronavirus) pandemic has had a huge impact on healthcare resources and staff in the UK. Understanding the key risk factors associated with infection amongst healthcare workers is essential for future pandemic response plans.

Currently there are scarce data relating to the infection rates and associated factors amongst healthcare workers in the United Kingdom (UK). Studies of infection rates in healthcare workers have largely relied on the real-time reverse transcriptase-polymerase chain reaction (RT-PCR) test to date and it appears that Healthcare workers are twice as likely to succumb to Coronavirus infection, when compared to the general population and those from Black and minority ethnic (BAME) backgrounds appear to be particularly at risk.

Currently there is no evidence that the presence of SARS-CoV-2 (severe acute respiratory syndrome coronavirus 2) antibodies provides seasonal or long term immunity to future infection.

Therefore, this study aims to understand the current level of SARS-CoV-2 antibody positivity and try to determine the likely risk to healthcare workers in the UK to COVID-19 infection. This study hopes to find out whether certain individual characteristics will have an impact on likelihood of infection susceptibility and antibody response and determine the impact of the presence of antibodies on the likelihood of future clinical infection over a 12 month period.

The study involves an initial online survey and linkage to the recent antibody test, then a further online survey in 6 and 12 months' time. The data obtained will be linked to data that the Human Resources Department (HR) holds.

Participants also have the option to partake in another antibody test at 6 and 12 months' time and linked to the data collected.

DETAILED DESCRIPTION:
Participants will have access to the study via the link given in an SMS (Short Message Service - text message) which will direct then to the first online survey.

They will then be contacted again in 6 and 12 months' time to complete the online survey again.

The survey answers will be linked to the results of the antibody tests by their mobile and Employment Number and also to data held about them by the HR Department.

The survey will take approximately 15 minutes to complete and will include questions on the following: profession; work-line type; demographics and behavioural factors; ethnicity; and symptoms (if COVID 19 was manifested).

Participants can also attend for another blood test (SARS-CoV-2 (severe acute respiratory syndrome coronavirus 2) antibody test) to detect any presence of antibodies at 6 and 12 months (optional) which will again be linked to the survey and HR data.

ELIGIBILITY:
Inclusion Criteria:

* All Staff employed by Royal Wolverhampton Trust, having undergone the SARS-CoV-2antibody test at the Trust's testing facility

Exclusion Criteria:

* Royal Wolverhampton NHS Trust staff who have not participated in antibody testing • Staff who have opted out to receiving the text message invite and be part of the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1504 (Actual)
Dates: Start 2020-11-24 (Actual); Primary Completion 2023-10-27 (Actual); Study Completion 2023-10-27 (Actual)

PRIMARY OUTCOMES:
The number of employees tested who have evidence of SARS-CoV-2 antibodies | 12 months
  evidence of SARS-CoV-2 antibodies
Factors associated with a positive test | 12 months
  Survey to establish
  * Type of healthcare role
  * Ethnicity
  * Age
  * Index of multiple deprivation
  * Previous RT-PCR test status
  * Previous clinical COVID infection
  * Previous period of self isolation
  * Level of COVID-19 related anxiety
  * Presence of one or more high risk factors for COVID 19
  * Presence or absence of self-reported COVID 19 symptoms
Likelihood of clinically relevant (causing illness) infection with SARS-CoV-2 in subjects with both positive and negative SARS-CoV-2 antibody tests | 12 months
  Infection compared to antibody presence

CONTACTS AND LOCATIONS:
Overall Officials: Supratik Basu, Principal Investigator — The Royal Wolverhampton NHS Trust
Locations (1):
- The Royal Wolverhampton NHS Trust, Wolverhampton, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Results will be published in journal

REFERENCES:
- [Result] Sethi S, Manuelpillai N, Mandal A, Simpson O, Morrissey H, Ball P, Sharrod-Cole H, Ford C, Whittaker AC, Drayson M, Race A, Bateman J, Basu S, Cotton J. COVID-19 seroprevalence after the first UK wave of the pandemic and its association with the physical and mental wellbeing of secondary care healthcare workers. Brain Behav Immun Health. 2022 Oct;24:100492. doi: 10.1016/j.bbih.2022.100492. Epub 2022 Aug 6. PMID 35957800